CLINICAL TRIAL: NCT05416281
Title: Customized Approaches for Evaluating and Reducing Chemical Exposures From Home Building Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00110402
Record Dates: First submitted 2022-06-05; First posted 2022-06-13 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-07

CONDITIONS: Environmental Exposure
Keywords: Environmental Exposure; Vacuum

STUDY DESIGN:
Intervention Model Description: Exposure will be evaluated before vacuuming and again after 8 weeks of vacuuming.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Vacuum Intervention (Experimental): This will include a home visit for environmental assessment AND a robotic vacuum intervention. Silicone wristbands will be used to evaluate exposure before and after a cleaning intervention.
  Interventions: Other: Robotic Vacuum
- No Intervention (No Intervention): This will include a home visit for environmental assessment.

INTERVENTIONS:
Other: Robotic Vacuum — Participants will be provided with a Roomba iRobot vacuum and will be asked to use the vacuum in their home for 8 weeks. Exposure to environmental exposures will be evaluated before and after the intervention using silicone wristbands.
  Arms: Robotic Vacuum Intervention

SUMMARY:
This project will evaluate new approaches to quantify and reduce chemical exposures from common building materials, with an emphasis on plastic additives, pesticides, flame retardants and lead in addition to other environmental contaminants. The objective of this project is to develop methods to quantify and reduce chemical exposures from the home environment using approaches that are adaptable and customizable to individuals and households. To achieve this goal investigators will: 1) Identify the types of building materials and housing characteristics associated with higher levels of exposure to different classes of contaminants; 2) Assess the effectiveness of a simple robotic vacuuming intervention for reducing exposure to a range of indoor contaminants; and 3) Evaluate a new wearable silicone wristband for monitoring exposure to lead and other metals.

DETAILED DESCRIPTION:
This study will leverage Project HOPE 1000 (Duke University Health System IRB Pro00100000), an existing longitudinal pregnancy cohort study. Investigators will invite a subset of women participating in HOPE 1000 (n=150) to participate in an environmental assessment involving home visits by a research team. Separate informed consent will be obtained from all participants. During home visits, environmental samples will be collected (e.g. dust and water) and participants will complete a questionnaire. A smaller subset of participants (n=50) will be asked to wear a silicone wristband to monitor ambient exposure to metals. Finally, to evaluate whether robotic vacuums can reduce exposure to environmental chemicals in the home, investigators will deploy robotic vacuum cleaners (i.e., Roomba) in 50 participants' homes. Investigators will measure a range of environmental contaminants and chemicals in environmental samples. This information will be combined with data and samples collected under the HOPE 1000 protocol. In particular, investigators will analyze maternal blood samples which have already been banked for metals and will analyze previously collected silicone wristbands for the same environmental chemicals targeted in previously collected samples.

Investigators will evaluate statistical associations between contaminants in the home and occupants' exposure. Investigators will also investigate changes in exposure before and after the intervention program. Risk to study participants includes the potential loss of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Participants enrolled in Project HOPE 1000, a pregnancy cohort study at Duke University Medical Center.
* Any enrolled HOPE 1000 participants planning to remain in their homes for at least the following 12 weeks will be eligible for our sub-studies.

Exclusion Criteria:

* Individuals not planning to remain in their homes for at least 12 weeks.
* Those not able to communicate in fluent English will be excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Change in Environmental Chemical Exposures | Participation will last through study completion, an average of 9 weeks
  Change in the mass of environmental chemicals on silicone wristbands will be evaluated after an 8-week vacuum intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Stapleton, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No